CLINICAL TRIAL: NCT07261761
Title: Cytokines as Diagnostic Markers of Pulpal Inflammation and Their Impact on the Outcome of Vital Pulp Therapy
Acronym: Pulp Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Khalifa, Researcher at faculty of dentistry Mansoura University, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M05060722
Record Dates: First submitted 2025-11-19; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2022-07

CONDITIONS: Reversible Pulpitis; Irreversible Pulpitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Molars or premolars with Reversible or irreversible pulpits (Experimental): fifteen patients with carious teeth showing signs and symptoms of pulp inflammation
  Interventions: Procedure: Vital pulp therapy; Procedure: blood sample collection
- Caries free molars or premolars (Active Comparator): fifteen patients with intact human premolars planed for extraction for orthodontic reason
  Interventions: Procedure: Extraction; Procedure: blood sample collection

INTERVENTIONS:
Procedure: Vital pulp therapy — 1. Full medical and dental history will be taken from each patient.
  2. Clinical and radiographic examination (Cone beam computed tomography) for the offending tooth.
  3. After anesthesia, Rubber dam is applied and complete caries removal will be done, deeply inside the cavity, the excavation will be done using low speed hand piece and excavator.
  4. A blood sample will be taken from the bleeding pulp tissue on a cotton pellet for Molecular test.
  5. After exposure, the pulp will be amputated to the level of the canal orifices (full pulpotomy) pulp vitality was confirmed by the presence of bleeding pulp tissue from all canals.
  6. Putty MTA will gently place over the pulp.
  7. The cavity will be sealed with initial deep layer of resin modified glass ionomer restoration (RMGI) and final superficial layer of composite restoration.
  Arms: Molars or premolars with Reversible or irreversible pulpits
Procedure: Extraction — 1. Full medical and dental history will be taken from each patient.
  2. Clinical and radiographic examination (Cone beam computed tomography) for the offending tooth.
  3. After anesthesia, Rubber dam is applied.
  4. A blood sample will be taken from the bleeding pulp tissue on a cotton pellet for Molecular test.
  5. Extraction for orthodontic reasons.
  Arms: Caries free molars or premolars
Procedure: blood sample collection — after access opening blood sample will be collected

SUMMARY:
intervention eligible patients with teeth diagnosed with reversible or irreversible pulpits will go for vital pulp therapy and the other group will be patients will go for extraction of caries free teeth for orthodontic reasons, blood samples will be collected from both groups to analyze the level of cytokines IL-8 and IL-10 and it's relation with the success of the pulp therapy

ELIGIBILITY:
Inclusion Criteria:

* The age ranges from 16-45 years medically free.
* Tooth should be vital on cold testing.
* Vital permanent premolar and molar on cold testing, with deep caries, subsequent pulp exposure and bleeding pulp tissue in all canals after complete pulpotomy.
* Diagnosis is either reversible or irreversible pulpitis with/ without periapical rarefaction.
* The tooth is restorable and free from advanced periodontal disease.
* Soft tissues around the tooth are normal with no swelling or sinus tract.

Exclusion Criteria:

* Patients over 45 years of age.
* Patients with clinical symptoms of periradicular inflammation or any periradicular radiographic lesions.
* Negative results for cold and electrical pulp testing

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Clinical success | one day, one, four and twelve weeks.
  post operative pain on cold testing binary outcome (Yes or no)

SECONDARY OUTCOMES:
Radiographic success | Pre-operative , and after six months
  Cone Beam Computed Tomography CBCT radiographic Examination for any periodontal widening or any periapical radiolucency.
level of cytokines | through study completion, an average of 6 months
  level of Interleukin 8 and Interleukin 10 will be measured using Enzyme- Linked Immunosorbent assay (ELISA) Kit

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura Univeristy, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided